CLINICAL TRIAL: NCT04633928
Title: Repair of Nasal Septal Perforations Using (Autologous) Nasal Chondrocyte Tissue Engineered Cartilage (N-TEC)- a Phase I Clinical Trial
Brief Title: Nasal Septum Perforation Treatment Using Tissue Engineered Cartilage Graft
Acronym: NSP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Dr Josef Vavrina, HNO Seepraxen, CH-8810 Horgen, Zurich (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02431
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Nasal Cartilage Septum Perforations
Keywords: Nasal chondrocytes; Nasal cartilage diseases; Septum perforation; Tissue engineering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-TEC (Experimental): N-TEC is based on autologous nasal chondrocytes expanded and further cultured on type I/III collagen membranes for about 2 weeks to allow cells to produce extracellular matrix containing cartilage specific proteins. The tissue engineered graft is then implanted in the nasal septum in an interposition graft with a temporoparietal fascia flap.
  Interventions: Biological: N-TEC: Autologous nasal chondrocytes and ECM proteins

INTERVENTIONS:
Biological: N-TEC: Autologous nasal chondrocytes and ECM proteins — Cells expanded in vitro and cultured in a collagen type I//III scaffold

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of implanting an engineered cartilage tissue in an interposition graft with a temporoparietal fascia (TPF) flap to repair medium size septal perforation. The engineered cartilage graft is obtained by culturing expanded autologous nasal chondrocytes within a collagen type I/III membrane. In addition, first data on efficacy will be collected.

DETAILED DESCRIPTION:
Nasal septum perforation (NSP) is a medical condition characterized by loss of cartilage and/or bony structures of the nasal septum together with their mucoperichondrium and mucoperiosteum. There are many causes for NSP like history of nasal surgery (iatrogenic), trauma, self-inflicted injuries, drugs, chemical irritants, neoplastic causes, inflammatory causes (vasculitides, Wegener's granulomatosis) or infections (syphilis, tuberculosis). The perforation in the nasal septum creates pathological turbulences in the nasal airflow, which result in a decrease of the normal humidification process. Depending on size and location of the defect, this can lead to serious discomfort for patients and reduction of their quality of life.

Since the current treatment methods (use of synthetic material, PDS, or of native cartilage) have disadvantages, the investigators want to show in a phase I study that the use of tissue engineered autologous nasal cartilage to repair perforations (holes) in the area of the nasal septum is suitable and safe. The engineered autologous nasal cartilage graft is used as a replacement for PDS or native cartilage in an interposition graft in the reconstruction of nasal septal perforations.

Before the operation, the subjective symptoms of the patients are recorded using two questionnaires: Nasal Obstruction Symptom Evaluation (NOSE) and Visual Analog Scale (VAS) and objective examinations are carried out with functional tests (rhinomanometry, acoustic rhinometry) and imaging (endoscopy, CT scans). A small biopsy taken from the nasal septum is processed in the laboratory, chondrocytes are isolated, expanded and cultured onto a collagen matrix to generate a tissue engineered cartilage graft. Subsequently, the engineered cartilage is implanted into the defect of the nasal septum. In the postoperative follow up at 6 weeks, 3, 6 and 12 months, the investigators examine whether the nasal septum is closed, the subjective symptoms of the patients are recorded and the objective measurements are carried out in order to compare them with the findings before the operation. The aim of the study is to show safety and feasibility and to gain initial data on effectiveness of this treatment (improvement of symptoms).

ELIGIBILITY:
Inclusion Criteria:

* • Nasal septal perforation of a medium size (diameter 0.5 to 2.0 cm), measured by endoscopy

  * Age above or equal to 18 years
  * Informed Consent as documented by signature
  * Patient is willing and able to give written informed consent to participate in the study and to comply with all study requirements, including attending all follow-up visits and assessments

Exclusion Criteria:

* • Nasal septal perforation of a small (<0.5 cm) or large size (>2.0 cm)

  * Patient is smoking
  * Known or suspected non-compliance, drug (especially cocaine) or alcohol abuse
  * Evidence of infection with HIV or hepatitis B or C, syphilis. Patients with a cured hepatitis B or C infection and/or verified antibodies are not excluded.
  * Known allergies to porcine collagen, penicillin or streptomycin
  * Women who are pregnant or breast feeding
  * Intention to become pregnant during the course of the study
  * Chronic treatment with steroids or immunomodulatory drugs
  * Diabetes
  * Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
  * Patient is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol or in a dependency or employment with the sponsor.
  * Patient is unable to understand the patient information
  * Patient has a known systemic connective tissue disease.
  * Patient has a known autoimmune disease.
  * Patient has a known immunological suppressive disorder or is taking immunosuppressive.
  * Patient is currently systemically or intra-articularly taking steroids and/or has used steroids within the 30 days prior to the planned treatment.
  * The patient has at the site of surgery an active systemic or local microbial infection, eczematization or inflammable skin alterations (including Protozoonosis: Babesiosis, Trypanosomiasis (e.g. Chagas-Disease), Leishmaniasis, persistent bacterial infections, such as Brucellosis, spotted and typhus fever, other Rickettsiosis, Leprosy, Recurrent Fever, Melioidosis or Tularaemia).
  * Patient has an active cancer.
  * Patient is currently participating, or has participated in any other clinical study within 3 months prior to the screening visit.
  * Patient has any other condition, which, in the opinion of the investigator, would make the patient unsuitable for the study.
  * Patient is unable to tolerate local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Safety assessment | one year follow up after implantation
  measured by reporting adverse events and reactions

CONTACTS AND LOCATIONS:
Overall Officials: Martin Haug, Prof, Principal Investigator — University Hospital Basel, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaiser B, Miot S, Wixmerten A, Pullig O, Eyrich M, Fulco I, Vavrina J, Schaefer DJ, Martin I, Barbero A, Haug MD. Engineered autologous nasal cartilage for repair of nasal septal perforations: a case series. Int J Surg. 2024 Oct 1;110(10):6573-6580. doi: 10.1097/JS9.0000000000001843. PMID 39197067